CLINICAL TRIAL: NCT01078181
Title: A Prospective Randomized Comparison on Weight Loss After Gastric Bypass and Banded Gastric Bypass Using the A.M.I B-Band (Soft Gastric Bypass Band)
Brief Title: Banded Versus Non-banded Roux-en-Y Gastric Bypass
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gerhard Prager / M.D., Medical University of Vienna / Department of Surgery
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUW ADIP STUDY 15; Banded Bypass Study 15 (Other: MUV - Metabolic and Bariatric Surgery)
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2009-11

CONDITIONS: Morbid Obesity
Keywords: gastric bypass; banded gastric bypass; weight loss; weight regain; bariatric surgery
MeSH Terms: conditions — Obesity, Morbid; Weight Loss | interventions — Gastric Bypass

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- banded gastric bypass (Active Comparator): Banded gastric bypass (circular anastomosis 21mm) using the A.M.I. B-Band (Soft Gastric Bypass Band)
  Interventions: Procedure: gastric bypass
- non-banded gastric bypass (Active Comparator): non-banded gastric bypass (circular anastomosis 21mm)
  Interventions: Procedure: gastric bypass

INTERVENTIONS:
Procedure: gastric bypass — laparoscopic gastric bypass with circular stapled 21mm gastrojejunostomy
  Other Names: laparoscopic gastric bypass; laparoscopic banded gastric bypass

SUMMARY:
This is a prospective randomized Study comparing Weight loss, Esophageal Motility and Reflux in lap. Gastric Bypass vs. lap. Banded-Gastric Bypass using the A.M.I. Soft Gastric Bypass Band (B-Band.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 40 or BMI > 35 + hypertension/diabetes mellitus
* pH metry and manometry preoperatively

Exclusion Criteria:

* formerly operations of the stomach
* formerly open abdominal surgery
* malignancy within the last 5 years
* formerly gastric banding

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-11; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Excessive Weight Loss | 3 years

SECONDARY OUTCOMES:
pouch dilatation, band migration, reflux, esophageal motility | 3 years
  Pouch dilatation verified by double contrast upper GI series Band migrations verified by gastroscopy Reflux verifies by pH-metry and gastroscopy Esophageal motility measured by manomerty

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Prager, M.D., Principal Investigator — Medical University of Vienna, Department of Surgery
Locations (1):
- Medical University of Vienna, Department of Surgery, Vienna, Austria